CLINICAL TRIAL: NCT03042533
Title: Union Rates of Transverse Tibia Fractures Managed With Internal Fracture Compression Through an Intramedullary Rod Compared to Standard Backslapping or Backslapping With Dynamic Locking
Brief Title: Union Rate of Transverse Tibia Fracture
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention. Low enrollment and PI leaving institution
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Claude Sagi, Professor, Orthopedics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001680
Record Dates: First submitted 2017-01-27; First posted 2017-02-03 (Estimated); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Closed Transverse Fracture of Shaft of Tibia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant Blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Conventional Compression (Active Comparator): Nail will be seated using conventional compression technique
  Interventions: Device: Conventional Compression
- Standard Backslapping (Active Comparator): Nail will be seated using standard backslapping technique
  Interventions: Device: Standard Backslapping
- Dynamic Locking with Backslapping (Active Comparator): Nail will be seated using backslapping with dynamic locking
  Interventions: Device: Dynamic Locking with Backslapping

INTERVENTIONS:
Device: Conventional Compression — Method of Nail fitting
  Arms: Conventional Compression
Device: Standard Backslapping — Method of Nail fitting
  Arms: Standard Backslapping
Device: Dynamic Locking with Backslapping — Method of Nail fitting
  Arms: Dynamic Locking with Backslapping

SUMMARY:
The investigators will compare the three methods of seating a tibial nail - Backslapping or Backslapping with Dynamic Locking or Internal Compression.

ELIGIBILITY:
Inclusion Criteria:

* Closed Tibia Shaft Fracture Treated with an IMN

Exclusion Criteria:

* Unable to consent due to language
* Unlikely to follow-up for one year

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Sagi, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Compression | Standard Backslapping | Dynamic Locking With Backslapping
Started | 1 | 4 | 1
Completed | 0 | 0 | 0
Not Completed | 1 | 4 | 1
Not completed — MD left program | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Compression | Standard Backslapping | Dynamic Locking With Backslapping | Total
Number analyzed (Participants) | 1 | 4 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 1 | 6
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 63 [63 to 63] | 37 [27 to 52] | 37 [37 to 37] | 42 [27 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 0 | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 4 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Healing of Tibia Fracture by Radiographic Exam
Description: Healing of Tibia Fracture by radiographic exam
Time Frame: One Year
Population: MD left institution project closed data not collected
Arm/Group | Conventional Compression | Standard Backslapping | Dynamic Locking With Backslapping
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 52 weeks
Arm/Group | Conventional Compression | Standard Backslapping | Dynamic Locking With Backslapping
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/4 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT03042533/Prot_SAP_000.pdf